CLINICAL TRIAL: NCT03691753
Title: Safety and Efficacy Study of Fitaya Vena Cava Filter for Deep Vein Thrombosis: A Multi-center, Randomized Controlled Trial
Brief Title: Safety and Efficacy Study of Fitaya Vena Cava Filter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT-01
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Venous Thromboembolism
Keywords: Fitaya; Vena cava filter
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Patients will be treated with Fitaya Vena Cava Filter System.
  Interventions: Device: Fitaya Vena Cava Filter System
- Control arm (Active Comparator): Patients will be treated with Aegisy Vena Cava Filter.
  Interventions: Device: Aegisy Vena Cava Filter

INTERVENTIONS:
Device: Fitaya Vena Cava Filter System — After the implantation of Fitaya Vena Cava Filter, the filter can be withdrawn from the patient within the window period (60 days) by using the withdraw system in junction of the sheath.
  Arms: Experimental arm
Device: Aegisy Vena Cava Filter — After the implantation of Aegisy Vena Cava Filter, the filter can be withdrawn from the patient within the window period (60 days) by using the withdraw system in junction of the sheath.
  Arms: Control arm

SUMMARY:
A Multi-center, Randomized Controlled Trial to evaluate the safety and efficacy of Fitaya Vena Cava Filter manufactured by Lifetech Scientific (Shenzhen) Co., LTD. for deep vein thrombosis.

DETAILED DESCRIPTION:
The trial was mainly for patients with high-risk deep vein thrombosis, and all subjects who passed the screening and signed the informed consent will be enrolled and be randomly divided into the experimental group and the control group according to the proportion of 1:1. For patients who will be allocated to the experimental group will be implanted with Fitaya Vena Cava Filters System, and for patients who will be allocated to the control group will be implanted with Aegisy Vena Cava Filters. Between 0 and 60 days, after the filter was implanted, the investigator will decide whether to withdraw the vena cava filter based on the subject's condition. If successfully withdraw the vena cava filter, the subject will be followed up for 1 month, if the withdraw is unsuccessful, the subject will be followed up for 180 days. This clinical trial is conducted in qualified clinical trial institutions with a planned duration of 16-24 months. Upon completion of the clinical trial report, it will be submitted together with other materials for the application for listing registration in the China Food and Drug Administration (CFDA).

ELIGIBILITY:
Inclusion Criteria:

1. Older or equal to 18 years of age, regardless of sex.
2. Patients are able to understand the purpose of the trial, voluntarily participated in and signed informed consent, and are willing to complete the follow-up as required by the program.
3. Patients diagnosed with inferior deep vein thrombosis (inferior vena cava, Iliac, femoral or popliteal DVT) or pulmonary embolism (PE), and concomitant with one or more of the following situation:

   1. with the existence of contraindications for anticoagulation therapy.
   2. complications such as bleeding occurred during anticoagulation therapy.
   3. pulmonary embolism still recurred after adequate anticoagulation therapy.
   4. All reasons cannot achieve sufficient anticoagulant.
   5. PE coexist with inferior DVT.
   6. Free thrombosis or large amounts of thrombosis are found in the iliac, femoral, popliteal or inferior vena cava.
   7. Patients with acute risk factors of DVT and PE needed to undergo abdominal, pelvic or lower limb surgery simultaneously.
   8. The patients had acute DVT, intend to do Catheter-Directed Thrombolysis (CDT, Percutaneous Mechanical Thrombectomy (PMT), or surgical thrombectomy.
4. The investigator determined that the patient had an appropriate femoral or jugular access for implantation of the filter.
5. The diameter of inferior vena cava intended to implant the filter is between 18mm and 29mm.

Exclusion Criteria:

1. Had been implanted with an inferior vena cava filter previously.
2. There is thromboembolism in the jugular or femoral vein access of the filter implantation.
3. Intended to permanently implant the filter.
4. Severe spinal deformity may affect the implantation or removal of filters.
5. Renal vein thrombosis, or, inferior vena cava thrombosis spread to renal vein.
6. Congenital malformation of inferior vena cava.
7. Having an uncontrolled infectious disease, such as bacteremia or toxaemia.
8. Active malignant tumour and tumour metastasis.
9. Allergic to imaging agents, materials of filters and conveyor (including nickel and titanium, polyester, Polytetrafluoroethylene (PTFE), nylon polymer materials).
10. Patients with X-ray contraindication.
11. Liver dysfunction: Alanine transaminase (ALT) or Aspartate transaminase (AST) was 2.5 times higher than the normal upper limit, Serum creatinine (Cr) was two times higher than the normal upper limit.
12. Abnormal coagulation function in patients: activated part of thrombin time (APTT)10s more than the normal value.
13. Patients with a life expectancy less than 12 months.
14. Patients with severe heart and lung dysfunction.
15. Pregnant or lactating, or woman planned to be pregnant.
16. The patients participated in clinical trials of other drugs or medical devices and did not come out of the group or withdraw within the first 3 months of the screening period of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-09-29 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The clinical success rate of the filter implantation | 6 months after implantation
  The clinically successful implantation of vena cava filter should meet the following three requirements simultaneously: 1. The filter was successfully implanted and the shape and positioning were satisfactory. 2. No symptomatic pulmonary embolism occurred in patients with permanent filter implantation within 6 months after implantation and was confirmed by Computed Tomography Pulmonary Angiography (CTPA). No symptomatic pulmonary embolism occurred in patients who had a removal of the filter during its indwelling and was confirmed by CTPA. 3. No rupture, no displacement, no venous penetration, no vena occlusion, no filter implantation or operation-related deaths occurred in the blood vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Zhang, Professor, Principal Investigator — Peking University People's Hospital
Locations (13):
- China (13):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Union Hospital Tongji College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Shandong University of TCM, Jinan, Shandong
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjing Medical University General Hospital, Tianjin, Tianjin Municipality
  - Frist Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang